CLINICAL TRIAL: NCT07133945
Title: Can the Number of Skin Tears be Reduced, by Prophylactic Treatment of the Skin in Dupuytrens Contracture Treated With Collagenase?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zealand University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: REG-185-2017
Record Dates: First submitted 2018-12-06; First posted 2025-08-21 (Actual); Last update posted 2025-08-21 (Actual); Status verified 2018-12

CONDITIONS: Dupuytren Disease of Finger
Keywords: Collagenase; Xiapex; Vaseline; Steristrip; Silicone
MeSH Terms: interventions — Petrolatum

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control group (No Intervention): This group will receive standard collagenase injection in the cord
- Experimental group (Experimental): This group will receive vaseline treatment, silicone plaster or steristrip on the skin overlying the cord before breakage of the cord
  Interventions: Procedure: Silicone plaster or Steristrip or Vaseline

INTERVENTIONS:
Procedure: Silicone plaster or Steristrip or Vaseline — Prophylatic treatment of the skin before breakage of the skin in dupuytrens disease
  Arms: Experimental group

SUMMARY:
Collagenase has gained pace in treating Dupuytrens contracture for some years. Thus this treatment is performed routinely in many orthopaedic and or hand surgical department. One of these benefits of the collagenase treatment is that the patients quickly recover and return to work or daily activities after the treatment. However, one of the often seen complications to the treatment is skin tear. This is reported in 20-80% of cases depending on the degree of contracture. The presence of skin tear leads to prolonged recovery, increased pain, scarring and post pone patients returning to daily activities and work. The investigators hypothesize that prophylactic initiatives with pre-existing products could reduce skin tear after treatment with collagenase injection into the Dupuytren cord.

DETAILED DESCRIPTION:
To the knowledge of the investigators no effective measures exists for preventing skin breakage following collagenase treatment of Dupuytrens disease. In the current study three different skin treatments are tested against a control group to see if skin breakage can be reduced by one of these prophylactic measures.

The study is performed as a prospective randomized non blinded study.

The degree of contraction is measured. Injection of collagenase into the cord. According to randomization the patient will be allocated to one of the following four treatments.

1. Standard treatment regime
2. Standard treatment regime + vaseline on skin over the cord and the hand is wrapped in a plastic glove till next day
3. Standard treatment regime + Silicone patch on skin over the cord and the hand is wrapped in a plastic glove till next day
4. Standard treatment regime + Steristrips on skin over the cord and the hand is wrapped in a plastic glove till next day

ELIGIBILITY:
Inclusion Criteria:

* Dupuytrens contracture
* Extension deficit of 30 degrees or more in the metacarpophangeal joint or the proximal interphalangeal joint

Exclusion Criteria:

* Previous treatment of the digit

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2018-06-30 (Actual); Study Completion 2018-06-30 (Actual)

PRIMARY OUTCOMES:
Tear of skin | During breaking af dupuytren cord following collagenase treatment. Time frame is thus within approximately 10 seconds
  Does the skin tear when breaking the dupuytren cord? yes or no. There is no recognized scale for this observation. Only the registration of the skin tearing or not.

CONTACTS AND LOCATIONS:
Locations (1):
- Zealand University Hospital, Køge, Region Sjælland, Denmark